CLINICAL TRIAL: NCT07126145
Title: Clinical Autoinflammatory Disease Cohort
Acronym: CAID
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Qiong Fu, Director, RenJi Hospital
Other Study IDs: LY2025-170-A
Record Dates: First submitted 2025-08-02; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Still Disease; Autoinflammatory Disease
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIDs patients: Patients with Still's disease must meet the 1992 Yamaguchi diagnostic criteria; patients with monogenic autoinflammatory diseases must meet the confirmed diagnostic criteria for the respective conditions; all patients must provide written informed consent.；Age range: 18-75 years old patients with autoinflammatory diseases.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — no interventions were involved

SUMMARY:
Autoinflammatory diseases (AIDs) are a group of rare disorders caused by dysregulation of the innate immune system, characterized by recurrent fever, systemic inflammation, and involvement of specific organs. Diagnosis relies on a combination of clinical features, laboratory tests, genetic findings, and response to treatment. Still's disease is a representative type of AID, marked by high spiking fevers, polyarthritis, evanescent rash, and markedly elevated inflammatory markers. Among its complications, macrophage activation syndrome (MAS) is the most life-threatening, affecting approximately 10-15% of patients. MAS involves uncontrolled immune activation and systemic inflammation, and if left untreated, may result in a mortality rate exceeding 50%. This study aims to develop a standardized clinical dataset and diagnostic-treatment framework for AIDs based on their disease characteristics. After establishing a data collection template, eligible patients aged 18-75 years with AIDs will be enrolled. Clinical data will be collected to build a prospective follow-up cohort, focusing particularly on adult-onset Still's disease (AOSD), to explore the clinical features and pathogenesis of AIDs.

DETAILED DESCRIPTION:
Autoinflammatory diseases (AIDs) are a group of rare disorders caused by overactivation of the body's innate immune system. They are marked by repeated episodes of fever, widespread inflammation, and damage to various organs. Because their symptoms can affect many different systems and often resemble other conditions, AIDs are frequently misdiagnosed or remain undetected for long periods.

The term "AIDs" covers more than 50 known single-gene (monogenic) diseases, as well as multi-gene (polygenic) conditions without an identified genetic cause. Examples include Still's disease, Behçet's disease, and certain types of inflammatory bowel disease. Adult-onset systemic autoinflammatory diseases (SAIDs) include Still's disease, Schnitzler syndrome, and idiopathic recurrent autoimmune pericarditis (IRAP). Common symptoms are periodic fevers of unknown origin, skin rashes, inflammation of membranes around organs (serositis), swollen lymph nodes, and joint pain or swelling. Laboratory findings often reveal elevated inflammatory markers such as ESR and CRP. These conditions can be further classified by their underlying pathways, including inflammasome-related diseases, type I interferonopathies, proteasome-related disorders, and NF-κB pathway-associated diseases.

Still's disease is a particularly rare type of SAID. It presents with high fevers, multiple joint pain, rash, and markedly increased inflammatory markers. The disease affects an estimated 2-6 people per million each year worldwide, but rates vary across populations. A serious complication, macrophage activation syndrome (MAS), develops in about 10-15% of patients. MAS involves uncontrolled immune activation and a massive release of inflammatory proteins known as cytokines-a process often called a "cytokine storm." Without rapid treatment, MAS can lead to multi-organ failure and has a mortality rate above 50%.

The exact cause of Still's disease and MAS remains unclear, but research shows it involves several intertwined processes: excessive immune cell activation, abnormal cytokine release, amplification of inflammation, and injury to multiple organs. Key inflammatory mediators include IL-1β, IL-6, IL-18, IFN-γ, and TNF-α. These molecules activate immune cells such as macrophages, neutrophils, and certain T cells, setting off a self-perpetuating cycle of inflammation. In addition, the formation of neutrophil extracellular traps (NETs) appears to play a role in tissue injury.

Because current diagnostic tools cannot reliably detect MAS early, and treatments-mainly glucocorticoids and immunosuppressants-are only partly effective and carry significant side effects, there is a pressing need for better understanding of the disease mechanisms. This study aims to follow a well-characterized cohort of patients with autoinflammatory diseases, particularly those with Still's disease and MAS, to identify new molecular targets and specific diagnostic biomarkers. The goal is to improve early detection, guide more precise treatments, and ultimately reduce mortality in these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adult-onset Still's disease (AOSD) according to the Yamaguchi criteria (as described above) or other established autoinflammatory disease diagnostic criteria.
* Age between 18 and 75 years, inclusive.
* Willingness and ability to comply with scheduled follow-up visits, examinations, and treatments.
* Voluntary provision of written informed consent.

Exclusion Criteria:

* Refusal or inability to provide informed consent; age under 18 or over 75 years; inability to provide at least 80% of the required core data for Still's disease or other autoinflammatory diseases.
* Presence of other connective tissue diseases.
* Positive detection of autoantibodies.
* Current acute infection or history of active tuberculosis.
* History of allergic constitution or multiple drug allergies.
* Psychiatric disorders or other conditions preventing compliance with examinations, follow-up, or treatment.
* Women who are currently pregnant or planning to become pregnant.
* Presence of malignant tumors.
* Participation in other clinical trials currently or within a specified washout period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18-75 years) diagnosed with autoinflammatory diseases.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Sustained Event-Free Remission | From the date of remission until the first documented disease progression, occurrence of treatment-related severe adverse events, or death from any cause, whichever occurred first, assessed up to 60 months.
  Proportion of participants who maintain clinical remission without experiencing disease-related complications or treatment-related adverse events, including glucocorticoid-associated toxicity.

SECONDARY OUTCOMES:
Glucocorticoid discontinuation rate | 3 months
  Proportion of patients who successfully taper and discontinue glucocorticoids
Time to biologic DMARD initiation | From enrollment to 36 months
  From enrollment to the start of biologic DMARD therapy
Time to first MAS event | From enrollment to 3 months
  Time from enrollment to first documented macrophage activation syndrome
Time to Onset of Glucocorticoid-Associated Complications | From initiation of glucocorticoid therapy to the first documented complication, with follow-up of up to 60 months.
  Time interval between the start of glucocorticoid treatment and the occurrence of the first treatment-related adverse event, including but not limited to infections, osteoporosis, hypertension, or diabetes.
Incidence of Treatment-Related Adverse Events | From treatment initiation to 36 months
  Number and proportion of participants who experience one or more adverse events attributable to treatment during the follow-up period. Adverse events may include infections, hepatic dysfunction, cytopenia, or other complications associated with immunosuppressants, glucocorticoids, or biologic agents.
Time to Relapse After Remission | From achievement of remission to first documented disease flare, with follow-up of up to 60 months.
  Duration between the time a participant first achieves clinical remission and the time of first subsequent disease relapse, defined by pre-specified clinical or laboratory criteria.